CLINICAL TRIAL: NCT02669641
Title: Complex Imaging Assessment of Steatosis in Patients Under Treatment With Combination Silimarin, Phyllanthus Niruri and Choline
Brief Title: Complex Imaging Assessment of Steatosis
Acronym: SteatoSPC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy Craiova (Other)
Collaborators: Fiterman Pharma SRL (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SteatoSPC; 1334/17.12.2015 (Other Grant/Funding Number: UMF Craiova)
Record Dates: First submitted 2016-01-23; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Fatty Liver
Keywords: Steatosis, Fatty liver, Steatohepatitis
MeSH Terms: conditions — Fatty Liver | interventions — Choline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Steatosis (Experimental): Patients with diagnosed steatosis in treatment with combination Silimarin, Phyllanthus Niruri and Choline
  Interventions: Dietary Supplement: Combination Silimarin, Phyllanthus niruri and Choline

INTERVENTIONS:
Dietary Supplement: Combination Silimarin, Phyllanthus niruri and Choline — Combination of one capsule: Phyllanthus niruri (225 mg), Silybum marianum (150 mg), Choline (60 mg) The dose: 3 capsules per day.
  Other Names: Stoptoxin Forte

SUMMARY:
The main objective is the assessment of MRI (Magnetic Resonance Imaging) Spectroscopy in patients diagnosed with hepatic steatosis in treatment with combination Silimarin, Phyllanthus Niruri and Choline.

DETAILED DESCRIPTION:
In the study will be included patients with alcoholic and non-alcoholic steatohepatitis evaluated in Research Center of Gastroenterology and Hepatology and Gastroenterology Clinic of University of Medicine and Pharmacy of Craiova. All the patients will undergo MRI and MRI Spectroscopy (3 Tesla) using PHILIPS INGENIA 3T System for exact steatosis quantification. The eligible patients will be treated with combination Silimarin, Phyllanthus Niruri and Choline (Stoptoxin Forte) for 6 months (in conformity Product Characteristics). After the treatment a new IRM Spectroscopy examination will be performed. All the acquired data will be analyzed and published.

ELIGIBILITY:
Inclusion Criteria:

* steatosis described on abdominal ultrasound

Exclusion Criteria:

* chronic viral hepatitis
* liver cancer
* abusive alcohol consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fat-fraction | 6 months after specific treatment
  MRI Spectroscopy is the most direct non-invasive MR-based method to separate the liver signal into its water and fat components and calculate a signal fat-fraction.
  To calculate the fat fraction record the area of lipid peak, the area of the water peak and the fat fraction is lipid area/(lipid area+ water area)×100.
  The signal fat-fraction with MRI Spectroscopy has a dynamic range of 0-100%. Steatosis grades are categorized into broad brackets of severity: grade 0 (normal) = up to 5% of cells affected, grade 1 (mild) = 5-33% of cells affected, grade 2 (moderate) = 34-66% of cells affected, and grade 3 (severe) ≥67% of cells affected.

CONTACTS AND LOCATIONS:
Overall Officials: Ioana Andreea Gheonea, Lecturer, Study Director — University of Medicine and Pharmacy Craiova
Locations (1):
- Research Center in Gastroenterology and Hepatology, University of Medicine and Pharmacy Craiova, Romania, Craiova, Please Select, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirpich IA, Miller ME, Cave MC, Joshi-Barve S, McClain CJ. Alcoholic Liver Disease: Update on the Role of Dietary Fat. Biomolecules. 2016 Jan 6;6(1):1. doi: 10.3390/biom6010001. PMID 26751488
- [Background] Gheonea DI, Saftoiu A, Ciurea T, Gorunescu F, Iordache S, Popescu GL, Belciug S, Gorunescu M, Sandulescu L. Real-time sono-elastography in the diagnosis of diffuse liver diseases. World J Gastroenterol. 2010 Apr 14;16(14):1720-6. doi: 10.3748/wjg.v16.i14.1720. PMID 20380003
- [Background] Bannas P, Kramer H, Hernando D, Agni R, Cunningham AM, Mandal R, Motosugi U, Sharma SD, Munoz del Rio A, Fernandez L, Reeder SB. Quantitative magnetic resonance imaging of hepatic steatosis: Validation in ex vivo human livers. Hepatology. 2015 Nov;62(5):1444-55. doi: 10.1002/hep.28012. Epub 2015 Sep 28. PMID 26224591